CLINICAL TRIAL: NCT02894606
Title: Influence of Thymoglobuline on Phenotypic and Functional Profiles of B Lymphocytes in Renal Transplant Recipients
Acronym: THYMO B
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: THYMO B (RB 13.072)
Record Dates: First submitted 2016-08-30; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Renal Transplant
Keywords: Kidney Transplant; Immunology

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood

GROUPS / COHORTS (2):
- Thymoglobulin Induction: Patient receiving thymoglobulin as an induction therapy for renal transplant
  Interventions: Drug: Thymoglobulin Induction
- Basiliximab Induction: Patient receiving basiliximab as an induction therapy for renal transplant
  Interventions: Drug: Basiliximab Induction

INTERVENTIONS:
Drug: Thymoglobulin Induction — The choice of the induction therapy is not a procedure of the study. This choice is made by the practioner, based on the graft recipient profile. This is a predefined group, the Thymoglobulin treatment is not an intervention in the study but must be considered as an exposure that is defined before the patient enters the study.
  Groups: Thymoglobulin Induction
Drug: Basiliximab Induction — The choice of the induction therapy is not a procedure of the study. This choice is made by the practioner, based on the graft recipient profile. This is a predefined group, the Basiliximab treatment is not an intervention in the study but must be considered as an exposure that is defined before the patient enters the study.
  Groups: Basiliximab Induction

SUMMARY:
The investigators expect to better characterise B cell subpopulation and functional properties early after graft, to analyse effect of induction therapy (thymoglobulin versus basiliximab) on B cells, and to compare this B cell profiles with those obtained in our previous study in patients with chronic Antibody Mediated Rejection (cAMR)

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Recipient of a renal allograft
* Patient receiving either basiliximab or thymoglobulin as in induction therapy for renal transplant
* Patient presenting a low immunologic risk
* Patient not opposed to his (her) study participation

Exclusion Criteria:

* Patient participating in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: kidney graft recipients from two French renal transplantation centers
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
The distribution of mature blood B cells subpopulations will be compared between the 2 groups | one year after renal transplant
Proliferation of freshly isolated cells T in presence of autologous B cells will be compared between the 2 groups. | one year after renal transplant

SECONDARY OUTCOMES:
Serum B-cell activating factor (BAFF) concentration comparison between the two groups | one year after renal transplant

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Le meur, Study Director — University Hospital, Brest
Locations (2):
- France (2):
  - CHU Brest, Brest
  - Tours University Hospital, Tours